CLINICAL TRIAL: NCT04821856
Title: A Randomized Placebo-controlled Trial of Cannabidiol to Treat Severe Behavioral Problems in Children and Adolescents With Intellectual Disability
Brief Title: Evaluation of the Effectiveness of Cannabidiol in Treating Severe Behavioural Problems in Children and Adolescents With Intellectual Disability
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Monash University (Other); University of Sydney (Other); Deakin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RCH HREC 70053
Record Dates: First submitted 2021-03-25; First posted 2021-03-30 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Intellectual Disability; Child Behavior Problem
Keywords: pediatric; intellectual disability; severe behavior problems
MeSH Terms: conditions — Intellectual Disability; Mental Disorders | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cannabidiol 100mg/ml (Experimental): The starting dose of cannabidiol (CBD) will be 5 mg/kg/day and will be administered orally twice daily in doses of 2.5 mg/kg (up titration phase from day 1 to 7). After one week, the dose of CBD will be increased to 10 mg/kg/day in two daily doses of 5mg/kg (8-week maintenance phase from day 8 to 63). On completion of the maintenance phase the dose of CBD will be decreased to 5mg/kg/day for one week (day 64 to 70), after which the CBD administration will cease.
  A ceiling dose of 1000mg/day will be administered to all participants weighing 100kg or greater. These participants will receive a dose of 500mg/day during up- and down-titration.
  Doses will be rounded to the nearest 10mg (0.1mL).
  Interventions: Drug: Cannabidiol Oil
- Placebo (Placebo Comparator): The control group will receive placebo medium-chain triglyceride (MCT) oil which is indistinguishable from the active medication in appearance, smell and taste.
  Dose will be matched for volume to the cannabidiol arm, and administered twice daily for 10 weeks (including up- and down-titration).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol Oil — Cannabidiol (CBD) isolate 100mg/ml in MCT oil oral solution, manufactured by THC Pharma
  Arms: Cannabidiol 100mg/ml
Drug: Placebo — MCT oil and flavoring solution, also manufactured by THC Pharma
  Arms: Placebo

SUMMARY:
This is a multi-site, double-blind, parallel group, randomized, placebo-controlled study of 140 participants comparing oral purified cannabidiol isolate (CBD) with placebo in reducing Severe Behavioral Problems (SBP) at 8 weeks in children aged 6 - 18 years with Intellectual Disability (ID). Eligible participants will be randomized 1:1 to receive either CBD or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 6 - 18 years of age;
2. DSM-5 diagnosis of intellectual disability (ID):

   1. Full scale IQ < 70 on standardized cognitive assessment. Testing results must be sighted by the investigators and performed within two years of enrollment. In the event that records of prior testing are unavailable or the assessment was more than 2 years prior, IQ will be estimated using the Wechsler Abbreviated Scale of Intelligence-II.
   2. Deficit in adaptive function (basis for severity rating of ID in DSM-5) in at least one activity of life on the Vineland Adaptive Behavior Scales (derives scores in Communication, Daily Living Skills and Socialization domains, and a Global Adaptive score). If records of prior testing are unavailable or the assessment was more than 2 years prior, this will be completed by the parent or guardian.
3. SBP: Defined as scores of:

   1. 18 or higher on the Aberrant Behavior Checklist-Irritability subscale (ABC-I), and
   2. moderate or higher on the Clinical Global Impressions-Severity scale;
4. No changes in either medication or other interventions in the 4 weeks prior to randomization, and intention to remain on same dose for the duration of the study;
5. Written informed consent from parent or legal guardian;
6. Participant and family have the ability to comply with the protocol requirements, in the opinion of the investigator.

Exclusion Criteria:

1. Non-English speaking parents;
2. Psychosis;
3. Taking clobazam, mTOR inhibitors (e.g sirolimus, tacrolimus), anti-cancer agents, citalopram >20mg/day, escitalopram >10mg/day.;
4. Abnormal liver function tests: defined as ALT > twice ULN;
5. Abnormal renal function tests: defined as creatinine > ULN
6. Current use of medicinal cannabis, or use in the 4 weeks prior to screening;
7. Pregnant or intending to become pregnant during the study, or breastfeeding;
8. Known allergy to cannabidiol or cannabis products

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 132 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
Mean difference between the cannabidiol 100mg/ml and placebo arms on the Aberrant Behavior Checklist-Irritability (ABC-I) subscale total score at day 64 | At day 64 (end of maintenance treatment period)
  This is a 15 item parent-rated questionnaire, used to measure Severe Behavioral Problems in children

SECONDARY OUTCOMES:
Mean difference between the cannabidiol 100mg/ml and placebo arms on the total scores of the four remaining subscales of the Aberrant Behavior Checklist (ABC) at day 64 | At day 64 (end of maintenance treatment period)
  43 parent-rated items assessing: Social withdrawal, Stereotypic behavior, Hyperactivity/Noncompliance and Inappropriate Speech
Comparison between the cannabidiol 100mg/ml and placebo arms of clinician ratings on the Clinical Global Impressions-Improvement at day 64. Data will be presented as the proportion of participants in each arm with a rating suggesting improvement | At day 64 (end of maintenance treatment period)
  This is a single item clinician-rated summary measure of improvement
Mean difference between the cannabidiol 100mg/ml and placebo arms on the total score of the Parent Rated Anxiety Scale-ASD at day 64 | At day 64 (end of maintenance treatment period)
  This is a 25 item parent-rated measure of anxiety in youth with ASD
Mean difference between the cannabidiol 100mg/ml and placebo arms on the total score of the Child & Adolescent Scale of Participation at day 64 | At day 64 (end of maintenance treatment period)
  This is a 20 item parent-rated questionnaire that includes sub-scales for participation in home, school, and community activities
Mean difference between the cannabidiol 100mg/ml and placebo arms on the weighted total score of the Child Health Utility 9D (CHU-9D) at day 64 | At day 64 (end of maintenance treatment period)
  This is a 9 item parent-rated, preference-weighted measure used to calculate quality adjusted life years for children
Mean difference between the cannabidiol 100mg/ml and placebo arms on the total score of the Sleep Disturbance Scale for Children at day 64 | At day 64 (end of maintenance treatment period)
  This is a 26 item parent-rated questionnaire assessing sleep difficulties in children
Mean difference between the cannabidiol 100mg/ml and placebo arms on the total score of the Assessment of Quality of Life 4D (AQOL-4D) at day 64 | At day 64 (end of maintenance treatment period)
  This is a 12 item self-report health-related instrument used to calculate quality adjusted life years for parents
Mean difference between the cannabidiol 100mg/ml and placebo arms on the total score of the Beach Center Family Quality of Life at day 64 | At day 64 (end of maintenance treatment period)
  This is a 25 item parent report measure that includes subscales assessing family interaction, parenting, emotional and material wellbeing, and disability-related support.
Mean difference between the cannabidiol 100mg/ml and placebo arms on the total score of the Depression Anxiety Stress Scale-21 at day 64 | At day 64 (end of maintenance treatment period)
  This is a 21 item self-rated assessment of parent mental health, including symptoms of depression, anxiety and stress
Mean difference between the cannabidiol 100mg/ml and placebo arms on the total score of the Autism Parenting Stress Index at day 64 | At day 64 (end of maintenance treatment period)
  This is a 13 item self-rated measure of 3 categories of stress drivers in parents: core social disability, difficult behavior, physical issues
The frequency of adverse events as reported on the modified version of the Liverpool Adverse Event Profile (LAEP) at day 64 will be summarised across the cannabidiol 100mg/ml and placebo arms | At day 64 (end of maintenance treatment period)
  Completed by the parent or guardian, the LAEP was designed to capture known side-effects of anti-epileptic medication. The modified version includes additional items to ascertain other known side-effects of CBD. This measure includes 34 items.

OTHER OUTCOMES:
Comparing the health sector cost-effectiveness of cannabidiol vs placebo in terms of Aberrant Behavior Checklist - Irritability (ABC-I) scores at day 64 | At day 64 (end of maintenance treatment period)
  This involves calculation of an incremental cost effectiveness ratio (ICER): health sector costs (CBD-placebo) divided by incremental ABC-I scores. Health sector costs will be calculated through: (1) Estimation of intervention costs from the study's financial records; (2) A brief Resource Use Questionnaire, completed by parents at day 64, which will capture medication and health sector resource use associated with their child's behaviour across the 8 week intervention period.
Comparing the societal cost-effectiveness of cannabidiol vs placebo in terms of Aberrant Behavior Checklist - Irritability (ABC-I) scores at day 64 | At day 64 (end of maintenance treatment period)
  This involves calculation of an incremental cost effectiveness ratio (ICER): societal costs (CBD-placebo) divided by incremental ABC-I scores. Societal costs will be calculated through a brief Resource Use Questionnaire, completed by parents at day 64, which will capture societal resource use and lost productivity associated with their child's behaviour across the 8 week intervention period.
Comparing the health sector cost-effectiveness of cannabidiol vs placebo in terms of Quality Adjusted Life Years calculated from the CHU-9D at day 64 | At day 64 (end of maintenance treatment period)
  This involves calculation of an incremental cost effectiveness ratio (ICER): health sector costs (CBD-placebo) divided by incremental Quality adjusted life years (QALYs) from CHU-9D . Health sector costs will be calculated through: (1) Estimation of intervention costs from the study's financial records; (2) A brief Resource Use Questionnaire, completed by parents at day 64, which will capture medication and health sector resource use associated with their child's behaviour across the 8 week intervention period.
Comparing the societal cost-effectiveness of cannabidiol vs placebo in terms of Quality Adjusted Life Years calculated from the CHU-9D at day 64 | At day 64 (end of maintenance treatment period)
  This involves calculation of an incremental cost effectiveness ratio (ICER): societal costs (CBD-placebo) divided by incremental Quality adjusted life years (QALYs) from CHU-9D . Societal costs will be calculated through a brief Resource Use Questionnaire, completed by parents at day 64, which will capture societal resource use and lost productivity associated with their child's behaviour across the 8 week intervention period.
Comparing the health sector cost-effectiveness of cannabidiol vs placebo in terms of Quality Adjusted Life Years calculated from the AQOL-4D at day 64 | At day 64 (end of maintenance treatment period)
  This involves calculation of an incremental cost effectiveness ratio (ICER): health sector costs (CBD-placebo) divided by incremental Quality adjusted life years (QALYs) from AQOL-4D . Health sector costs will be calculated through: (1) Estimation of intervention costs from the study's financial records; (2) A brief Resource Use Questionnaire, completed by parents at day 64, which will capture medication and health sector resource use associated with their child's behaviour across the 8 week intervention period.
Comparing the societal cost-effectiveness of cannabidiol vs placebo in terms of Quality Adjusted Life Years calculated from the AQOL-4D at day 64 | At day 64 (end of maintenance treatment period)
  This involves calculation of an incremental cost effectiveness ratio (ICER): societal costs (CBD-placebo) divided by incremental Quality adjusted life years (QALYs) from AQOL-4D . Societal costs will be calculated through a brief Resource Use Questionnaire, completed by parents at day 64, which will capture societal resource use and lost productivity associated with their child's behaviour across the 8 week intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Daryl Efron, Study Director — Murdoch Childrens Research Institute
Locations (3):
- Australia (3):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Monash Children's Hospital, Clayton, Victoria
  - Royal Children's Hospital / Murdoch Children's Research Institute, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set collected for this analysis of the RCT of CBD in children and adolescents with ID will be available six months after publication of the primary outcome. The study protocol and analysis plan will also be available. The data must be obtained from the Murdoch Children's Research Institute. Prior to releasing any data the following are required: a data access agreement must be signed between relevant parties, the 'RCT of CBD in children and adolescents with ID' Trial Steering Committee must see and approve the data analysis plan describing how the data will be analysed, there must be an agreement around appropriate acknowledgment and any additional costs involved must be covered. Should the Trial Steering Committee be unavailable, this role is delegated to the Murdoch Children's Research Institute. Data will only be shared with a recognized research organisation which has approved the proposed analysis plan.
Supporting Information: Study Protocol, SAP
Time Frame: 6 months after publication of primary outcome
Access Criteria: 1) Data access agreement; 2) approval by Trial Steering Committee; 3) recognized research institutions.

REFERENCES:
- [Background] Efron D, Taylor K, Payne JM, Freeman JL, Cranswick N, Mulraney M, Prakash C, Lee KJ, Williams K. Does cannabidiol reduce severe behavioural problems in children with intellectual disability? Study protocol for a pilot single-site phase I/II randomised placebo controlled trial. BMJ Open. 2020 Mar 8;10(3):e034362. doi: 10.1136/bmjopen-2019-034362. PMID 32152170
- [Background] Efron D, Freeman JL, Cranswick N, Payne JM, Mulraney M, Prakash C, Lee KJ, Taylor K, Williams K. A pilot randomised placebo-controlled trial of cannabidiol to reduce severe behavioural problems in children and adolescents with intellectual disability. Br J Clin Pharmacol. 2021 Feb;87(2):436-446. doi: 10.1111/bcp.14399. Epub 2020 Jul 1. PMID 32478863